CLINICAL TRIAL: NCT06881628
Title: Efficacy of Tranexamic Acid and Vitamin k Injection in Control of Upper Gastrointestinal Bleeding in Egyptian Cirrhotic Patients: A Randomized Controlled Study
Brief Title: Tranxemic Acid and Vitamin K Injection to Control Upper Gastrointestinal Bleeding in Cirrhotic Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Rania Mamdouh Elkafoury, Lecturer of Tropical Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36264PR982/12/24
Record Dates: First submitted 2025-03-04; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Upper Gastrointestinal Bleeding (UGIB); Variceal Bleeding; Cirrhosis
Keywords: Variceal bleeding; Tranexamic acid and vitamin K; Liver cirrhosis
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Fibrosis; Liver Cirrhosis | interventions — Tranexamic Acid; Vitamin K

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tranexamic acid and vitamin K (Experimental): 97 cirrhotic patients presenting with UGIB receiving tranexamic acid (1 g loading dose followed by 3 g maintenance dose over 24-48 hours) and intravenous injection of 10 mg daily of vitamin K for 24-48 h. Intervention will be carried out besides the recommended initial management of airway management, hemodynamic stabilization, octreotide analogue, PPI, antibiotics, and endoscopy.
  Interventions: Drug: Tranexamic Acid and vitamin K
- Placebo (Placebo Comparator): 97 cirrhotic patients presenting with UGIB receiving IV saline besides the recommended initial management of airway management, hemodynamic stabilization, octreotide analogue, PPI, antibiotics, and endoscopy.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid and vitamin K — Tranxemic acid (1 g loading dose followed by 3 g maintenance dose over 24- 48 hours) and intravenous injection (10 mg daily of vitamin K for 24-48 h) along with initial management of airway management, hemodynamic stabilization, octreotide analogue, PPI, antibiotics, and endoscopy to control UGIB in cirrhotic patients.
  Patients will be followed up after 5 days and 6 weeks to assess the rate of rebleeding, need for blood transfusion, hospital stay, adverse effects, and mortality rate.
  Arms: Tranexamic acid and vitamin K
Drug: Placebo — Intravenous saline over 24-48 hours along with initial management of airway management, hemodynamic stabilization, octreotide analogue, PPI, antibiotics, and endoscopy to control UGIB in cirrhotic patients.
  Patients will be followed up after 5 days and 6 weeks to assess the rate of rebleeding, need for blood transfusion, hospital stay, adverse effects, and mortality rate.
  Arms: Placebo

SUMMARY:
The goal of this randomized controlled clinical trial is to evaluate the efficacy of Tranexamic acid and vitamin K injection versus placebo in control of upper gastrointestinal bleeding (UGIB) in Egyptian cirrhotic patients.

Researchers will compare the bleeding and mortality rates (at 5 days and 6 weeks post endoscopic intervention for UGIB) between patients receiving tranxemic acid and vitamin K injection and patients receiving placebo.

Participants presenting with variceal bleeding will be randomly assigned to receive tranexamic acid (1 g loading dose followed by 3 g maintenance dose over 24- 48 hours) and intravenous injection of 10 mg daily of vitamin K for 24-48 h or matching placebo group receiving IV saline. Intervention will be carried out besides the recommended initial management of airway management, hemodynamic stabilization, octreotide analogue, PPI, antibiotics, and endoscopy.

Follow-up All patients will be kept at the hospital for at least 5 days from the index bleed and will be discharged if no other reason was observed to keep them at the hospital.

The rate of rebleeding, need for blood transfusion, hospital stay, adverse effects, and mortality rate were evaluated and compared across the groups.

At discharge, all patients will be started on nonselective beta-blockers if there was no contraindication. They will be given instructions to attend to hospital if they noticed any melena or hematemesis.

Second follow-up after 6 weeks for the rebleeding rate and mortality related to bleeding rate.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Liver cirrhosis
* Upper gastrointestinal bleeding

Exclusion Criteria:

* Patients aged < 18 years
* Allergy to tranexamic acid
* Allergy to vitamin K injection
* DIC.
* Thromboembolic event.
* Pregnancy or lactation.
* End-stage renal disease.
* Unwilling to participate in our study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Rebleeding rate | through study completion, an average of 1 year
  The rate of rebleeding and need for blood transfusion at 5 days and 6 weeks will be evaluated and compared across the groups.

SECONDARY OUTCOMES:
Mortality rate | through study completion, an average of 1 year
  The mortality rates at 5 days and 6 weeks will be evaluated and compared across the groups.
adverse effects | through study completion, an average of 1 year
  Drug adverse effects at 5 days and 6 weeks will be evaluated and compared across the groups.

CONTACTS AND LOCATIONS:
Overall Officials: Rania M Elkafoury, MD, Principal Investigator — Tropical medicine and infectious diseases Department, Faculty of Medicine, Tanta University
Locations (1):
- Tanta University Hospitals, Tanta, Gharbyea, Egypt